CLINICAL TRIAL: NCT01625481
Title: Prospective, Single Arm, Open Label, Non-randomized Study to Evaluate The Safety and Performance of The Seal-V System
Brief Title: Seal-V Safety and Performance Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sealantis Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WP2-072-02
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: C.Surgical Procedure; Vascular (Peripheral)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Seal-V (Experimental): A vascular sealant intended to achieve adjunctive hemostasis by mechanically sealing areas of potential leakage in surgical reconstruction of large blood vessels.
  Interventions: Device: Seal-V

INTERVENTIONS:
Device: Seal-V — Seal-V is applied adjunctively to cover the suture lines.
  Other Names: SEAlantis Vascular WP2(A)

SUMMARY:
The purpose of this study is to further assess the safety and performance of Seal-V as an adjunct to standard surgical procedure for achieving hemostasis in patients undergoing peripheral vascular reconstruction surgeries using synthetic grafts.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of >18 years of age
* Signed Informed Consent
* Patients requiring vascular reconstruction surgeries using synthetic (such as PTFE, Dacron) or autologous (such as native veins) grafts, including the following:
* Peripheral bypass surgeries, such as arterio-arterial bypasses [including: axillo-(bi)femoral, ilio-(bi)femoral, femoro-femoral, ilio-popliteal, femoro-popliteal (including below knee), femoro-tibial vessel bypass]
* Arteriovenous (AV) dialysis access shunt in the upper or lower extremity
* Patients able and willing to complete all follow-up visits

Exclusion Criteria:

* Vascular surgery other than peripheral bypass surgeries and arteriovenous (AV) dialysis access shunt procedures as described above
* Reoperation at the same treatment site
* Known sensitivity to device materials, such as indigo carmine dye or alginate
* Pregnant or lactating women
* Systemic infection
* Participation in another clinical trial or treatment with any investigational agent in past 30 days
* Congenital coagulation disorders (e.g., thrombocytopenia [<100,000 platelet count], thromboasthenia, hemophilia, or von Willebrand disease)
* Severe congenital or acquired immunodeficiency (e.g., HIV infection or long term treatment with immunosuppressive drugs)
* Prior radiation therapy to the operating field

Intraoperative Exclusion Criteria:

* Major intraoperative complications that require resuscitation or deviation from the planned surgical procedure
* Intraoperative change in planned surgical procedure that results in the patient no longer meeting preoperative inclusion and/or exclusion criteria
* Local infection at the operating field

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-07; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
TTH, Time to Hemostasis | Perioperative; within 10 minutes after clamp release
  Duration from the point at which circulation is restored to the graft/artery until bleeding ceases at the treatment site

SECONDARY OUTCOMES:
Successful cessation of bleeding at a treatment site | Perioperative; within 10 minutes after clamp release
Intraoperative blood loss | Perioperative
  Measured by weighing the surgical swabs used only in the application area and used from the time Seal-V was applied until hemostasis
Incidence of successful deployment of the Seal-V device | Perioperative

CONTACTS AND LOCATIONS:
Overall Officials: Rina Lev, PhD, Study Director — Sealantis Ltd.
Locations (3):
- Israel (3):
  - Department of Vascular Surgery, Bnai-Zion Medical Center, Haifa
  - Vascular Surgery Department, Rambam Health Care, Haifa
  - Department of Vascular Surgery, Chaim Sheba Medical Center, Tel Litwinsky